CLINICAL TRIAL: NCT05365568
Title: Left Bundle Branch Area Pacing Using Conventional Stylet Driven Pacemaker Leads for Cardiac Resynchronization Therapy: a Randomized Study
Brief Title: Left Bundle Branch Area Pacing Using Conventional Stylet-driven Pacemaker Leads for Cardiac Resynchronization Therapy
Acronym: LeCaRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jean-Benoît Le Polain de Waroux, Coordinating Principal Investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LeCaRT
Record Dates: First submitted 2022-04-29; First posted 2022-05-09 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure with Reduced Ejection Fraction
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LBBAP (Experimental)
  Interventions: Procedure: Left Bundle Branch Area Pacing (LBBAP)
- BiV (Active Comparator)
  Interventions: Procedure: Biventricular pacing (BiV)

INTERVENTIONS:
Procedure: Left Bundle Branch Area Pacing (LBBAP) — Left bundle branch area pacing using conventional stylet driven pacemaker leads for cardiac resynchronization therapy
  Arms: LBBAP
Procedure: Biventricular pacing (BiV) — Cardiac resynchronization therapy (CRT) using biventricular pacing (BiV)
  Arms: BiV

SUMMARY:
The aim of this study proposal is to compare the effectiveness of two distinct pacing modalities for cardiac resynchronization therapy. Our primary hypothesis is that left bundle branch area pacing (LBBAP) using conventional stylet driven pacemaker leads is an effective resynchronization method that yield to at least similar clinical benefits and outcomes when compare to biventricular pacing.

DETAILED DESCRIPTION:
Recently some retrospective or uncontrolled studies were published that compared cardiac resynchronization therapy (CRT) using left bundle branch area pacing (LBBAP) and biventricular pacing (BiV), although with a limited number of patients. Moreover, only one of these studies compared LBBAP + right ventricle stimulation to conventional BiV stimulation prospectively. None of the studies used conventional stylet-driven pacemaker leads for LBBAP. Therefore, the present trial aims to fill-in the gap in the current literature regarding LBBAP for CRT and provide a first randomized head-to-head comparison against CRT.

The aim of this study proposal is to compare the effectiveness of two distinct pacing modalities for cardiac resynchronization therapy. Our primary hypothesis is that left bundle branch area pacing (LBBAP) using conventional stylet driven pacemaker leads is an effective resynchronization method that yields to at least similar clinical benefits and outcomes when compared to biventricular pacing.

The study is a multicentre, randomized trial comparing LBBAP against biventricular pacing. After characterization of the type device implanted (Pacing or Defibrillator), randomization will occur between both groups in a 1:1 ratio. The trial purpose is to demonstrate the efficacy of LBBAP to treat clinical heart failure in-patient indicated to receive a CRT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Left Ventricular Ejection Fraction (LVEF) and NYHA meeting one off the previous indications documented with transthoracic echocardiography (TTE) no later than 3 months before randomization.
* New York Heart Association (NYHA) class II-IV
* Baseline left bundle branch block and QRS &gt;130ms or QRS &gt;150ms of any morphology or a wide paced QRS duration.

Exclusion Criteria:

* Younger than 18 years old
* Pregnancy
* Any unstable medical condition, life expectancy &lt; 12 months
* Inability to provide consent or to undergo follow-up
* Narrow QRS duration (≤130ms) or prolonged QRS duration with typical Right Bundle Branch Block (RBBB) morphology on 12 lead ECG and sinus rhythm.
* Significant hypertrophic cardiomyopathy - any septum abnormality contra-indicating LBBAP implantation (according to physician's evaluation)
* Patients who are unable to perform a 6 minute walk test (6MWT) Note: patients should be able to perform a 6 minute walk test, but it is not a requirement to have the test performed before the procedure (e.g. due to inability of planning).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of days elapsed from study procedure to first occurrence of one of the following events (combined endpoint) or to study close-out in the total patient population. | 12 months
  First occurrence of one of the following clinical events: death, hospitalization or unscheduled visit for heart failure (HF) or worsening HF symptoms with adaptation of the medical therapy, implant failure for any cause, implantable electronic cardiac device (IECD) re-intervention for any reason during follow-up (Lead Dislocation/phrenic nerve stimulation…)

SECONDARY OUTCOMES:
Improvement of procedural characteristics: Operative and fluoroscopic times | 1 day
  Improvement of procedural characteristics: Operative and fluoroscopic times
Correction of electrical desynchrony post-implant | 1/6/12 months
  Correction of electrical desynchrony post-implant, at 1/6/12 months
Clinical functional response (6MWT) | 6 months
  Clinical functional response as evaluated by the improvement of the 6 Minutes Walk Test (6MWT) at 6 months follow-up
Left ventricular reverse remodelling | 6/12 months
  Left ventricular reverse remodelling at 6 and 12 months follow-up as evaluated by the reduction of the Left Ventricular End-systolic Volume (LVESV) using trans-thoracal echocardiography
Implantable cardioverter defibrillator (ICD) therapies | 6/12 months
  ICD therapies at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Benoît le Polain de Waroux, MD, PhD, Principal Investigator — AZ Sint Jan Brugge AV
Locations (11):
- Belgium (11):
  - UZA, Edegem, Antwerpen
  - CHU Charleroi, Lodelinsart, Henegouwen
  - Jessa Ziekenhuis Hasselt, Hasselt, Limburg
  - CHR Citadelle Liège, Liège, Liège
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - UCL Saint-Luc, Woluwe-Saint-Lambert, Vlaams-Brabant
  - Clinique Saint-Pierre Ottignies, Ottignies-Louvain-la-Neuve, Waals-Brabant
  - AZ Sint-Jan Brugge, Bruges, West-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen
  - CHU HELORA - Site Jolimont, Haine-Saint-Paul

IPD SHARING:
Plan to Share IPD: No